CLINICAL TRIAL: NCT01102829
Title: Early Migration in a High Congruent Rotating Platform Total Knee Prosthesis Design. A Synchronised Motion Analysis Study With Fluoroscopy and RSA
Brief Title: Early Migration in a High Congruent Rotating Platform Total Knee Prosthesis Design
Acronym: ROCC
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: N. Wolterbeek, MSc (principal investigator), Leiden University Medical Center
Other Study IDs: ROCC
Record Dates: First submitted 2010-04-09; First posted 2010-04-13 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Knee Joint; Arthroplasty; Replacement; Knee
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to accurately assess the relationship between knee joint kinematics and migration of the tibial component of a high congruent, rotating platform total knee prosthesis by using fluoroscopy synchronised in time and space with a force plate, an external motion registration system and Electromyography (EMG).

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with osteoarthritis and requiring primary arthroplasty
* Patient is capable of giving informed consent and expressing a willingness to comply with this study
* Patient has no major deformities
* The ability to perform a lunge and step-up motion without the help of bars or a cane.
* No or slight pain during activity according to the Knee Society Pain Score (Ewald, 1989; Insall et al., 1989)

Exclusion Criteria:

* The patient is unable or unwilling to sign the Informed Consent specific to this study
* The individual has a functional impairment of any other lower extremity joint besides the operated knee
* Patient has a flexion contracture of more than 15°
* Patient has a varus/valgus contracture of more than 15°
* Patients requiring revision arthroplasty
* The patient does not understand the Dutch or English language good enough to participate.
* The use of walking aids
* The inability to walk more than 500 meters

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2007-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Migration | 24 months post-operatively
  Roentgen stereophotogrammetric analysis is used to determine the migration of the prosthesis with respect to the bone.

SECONDARY OUTCOMES:
anterior-posterior translation patterns | 6 months post-operatively
  Fluoroscopy was used to determine the anterior-posterior translation patterns of the femoral component with respect to the tibial component.
Axial rotation patterns | 6 months post-operatively
  Fluoroscopy was used to determine the axial rotation patterns of both the insert and the femoral component with respect to the tibial component
Muscle activity | 6 months post-operatively
  Bipolar surface EMG data of the flexor and extensor muscles is collected.
Shear forces | 6 months post-operatively
  A force plate is used to measure the ground reaction forces which can be used to calculate the shear forces.

CONTACTS AND LOCATIONS:
Overall Officials: Rob GH Nelissen, Prof, MD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands